CLINICAL TRIAL: NCT02912247
Title: A Open, Randomized, Single-dose, Comparative Bioequivalency and Safety Study of Human Recombinant Anti-tumor Necrosis Factor Alpha Monoclonal Antibody Injection and Adalimumab in Chinese Healthy Volunteers
Brief Title: Comparative Clinical Trial to Evaluate Bioequivalency and Safety of Monoclonal Antibody Injection and Adalimumab in Chinese Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIBI303A201
Record Dates: First submitted 2016-09-21; First posted 2016-09-23 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2018-06

CONDITIONS: Healthy
Keywords: tumor necrosis factor-a blocker; pharmacokinetics; safety
MeSH Terms: interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- monoclonal antibody injection (Experimental): human recombinant anti-tumor necrosis factor alpha monoclonal antibody injection 40mg administered subcutaneously once
  Interventions: Drug: human recombinant anti-tumor necrosis factor alpha monoclonal antibody injection
- adalimumab (Active Comparator): adalimumab 40mg administered subcutaneously once
  Interventions: Drug: adalimumab

INTERVENTIONS:
Drug: human recombinant anti-tumor necrosis factor alpha monoclonal antibody injection — human recombinant anti-tumor necrosis factor alpha monoclonal antibody injection, 40mg,subcutaneous injection,once
  Arms: monoclonal antibody injection
Drug: adalimumab — adalimumab, 40mg,subcutaneous injection,once
  Arms: adalimumab

SUMMARY:
This clinical study is a phase 1 study which carried out to establish the pharmacokinetic equivalence and equal safety of human recombinant anti-tumor necrosis factor alpha monoclonal antibody injection and Adalimumab when used as a single subcutaneous injection in healthy volunteers.

DETAILED DESCRIPTION:
This is a comparative, open, randomized clinical study. The purpose of the study is to demonstrate that human recombinant anti-tumor necrosis factor alpha monoclonal antibody injection is equivalent to adalimumab in terms of pharmacokinetics and safety after single subcutaneous injection in Chinese healthy volunteers.The study will enroll 180 healthy volunteers, who will be randomized into 2 groups.

ELIGIBILITY:
Inclusion Criteria:

1. Male, age between 18 and 55;
2. Body weight≥50kg and body mass index(BMI) within the range 19 to 28 kg/m2;
3. To fully understanding the purpose of the study, to understand the pharmacological action of the study drugs and the possible adverse reactions; participants who are voluntary to sign the informed consent according to the Declaration of Helsinki.

Exclusion Criteria:

1. History of adalimumab treatment;
2. History of relevant allergy/hypersensitivity(including allergy to the study drug or its ingredient );
3. Participation in another interventional trial within 3 months prior to administration of the study drug;
4. Blood donation(more than 200 mL within 12 weeks prior to administration of the study drug);
5. Use of any drugs(including traditional Chinese medicine) within 2 weeks or at least 5 half-lives(whichever is longer) prior to administration;
6. History of cluster of differentiation 4 antagonist or tumor necrosis factor alpha antagonist use, or use tumor necrosis factor antagonist(such as thalidomide) 3 months prior to administration;
7. Abnormal significant clinically chest radiograph, ECG, or laboratory examinations at screening and Baseline, judged by the investigators;
8. History of opportunistic infection(s)(such as: herpes zoster, mycoplasma, Pneumocystis carinii, histoplasma, Aspergillus, mycobacterium) within 6 months prior to screening;
9. Known recurrent or chronic infectious disease(s) history, including but not limited to: chronic kidney infect, chronic chest infection(such as bronchiectasis), nasosinusitis, recurrent urinary tract infection, open, drainage or infected wounds of the skin;
10. Tuberculosis(TB) history, or suspected clinically TB(including but not limited to: pulmonary tuberculosis, lymphoid tuberculosis, tuberculous pleurisy), or a positive Tuberculosis spot test;
11. Positive serology for human immunodeficiency virus(HIV) antibody;
12. Positive serology for hepatitis C virus antibody;
13. Active or chronic hepatitis B virus infection, such as positive hepatitis B virus surface antigen;
14. History of organ transplant(except for corneal transplantation≥3 months prior to Screening);
15. Known immunodeficiency history;
16. Use a live vaccine within 3 months prior to administration;
17. Alcohol or drug abuse within 12 months prior to Screening; unwilling/inability to refrain from alcohol from 72 hours prior to administration and until during the trial period;
18. Unwilling to use adequate contraception(such as condoms) during the study period;
19. Evidence suggests presence of clinically significant hepatic, renal, gastrointestinal, cardiovascular, endocrine, respiratory, hematologic, or neurologic abnormality;
20. Mentally impaired;
21. Disabilities, bed rest, wheelchair dependent, or lack of activity of daily life;
22. Subjects who are unsuited to the study for any reason, judged by the investigators.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 183 (Actual)
Dates: Start 2016-10-27 (Actual); Primary Completion 2017-09-22 (Actual); Study Completion 2017-09-22 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve from time zero to the last quantifiable concentration(AUClast) | 71days
Area under the concentration-time curve from time zero to infinity(AUCinf) | 71days
Maximum serum concentration(Cmax) | 71days

SECONDARY OUTCOMES:
Time to reach the maximum concentration(Tmax) | 71days
Elimination rate constant(γz) | 71days
Terminal half-live(T1/2) | 71days
Apparent clearance(CL/F) | 71days
Apparent volume of distribution(V/F) | 71days

CONTACTS AND LOCATIONS:
Overall Officials: Bei Hu, Professor, Principal Investigator — Peking Union Medical College Hospital

IPD SHARING:
Plan to Share IPD: No